CLINICAL TRIAL: NCT01718171
Title: Progression of the Systemic Inflammatory Response in Patients With Appendicitis
Brief Title: Inflammatory Response in Appendicitis
Status: Completed | Type: Observational
Sponsor: Cirujanos la Serena (Other)
Responsible Party: Principal Investigator, MARCELO A. BELTRAN, M.D., DIGESTIVE SURGEON, Cirujanos la Serena
Other Study IDs: HLS-0044-2012
Record Dates: First submitted 2012-10-29; First posted 2012-10-31 (Estimated); Last update posted 2012-10-31 (Estimated); Status verified 2012-10

CONDITIONS: Appendicitis
Keywords: Appendicitis; SIRS; C-reactive protein
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group I, Group II, Group III, Group IV: Values and results of the Systemic Inflammatory Response and C-reactive protein to appendicitis

SUMMARY:
Although the presence of SIRS has been described in patients with appendicitis, its progressive response related and together with progression of symptomatology from the onset of symptoms to diagnostic has not been characterized. Continuation of the systemic inflammation in patients with injury and infectious processes may result in multiple organ dysfunction and ultimately failure. As with any acute inflammatory condition, the patients' systemic inflammatory response to appendicitis will progress and become more intense with the passing of time. The purpose of this study is to characterize the systemic inflammatory response to appendicitis from the beginning of symptoms to diagnostic in patients with appendicitis submitted to emergency surgery.

DETAILED DESCRIPTION:
* A prospective non-interventional, observational, descriptive study was conducted.
* At our institution a median of 250 adult patients are submitted to emergency appendectomy every year. From this universe, a sample of 152 patients with a power of 80%, an error of 5% and 95% Confidence Intervals was required to perform this study.
* We included 268 patients in the database, of them 85 cases that did not comply with the inclusion criteria were excluded from the analysis. A total of 183 patients (100%) selected according to the following criteria were studied: Patients with appendicitis confirmed by histology operated on our institutional Emergency Unit with an age range from 15 to 80 years.
* Any patient with immunosuppressive or immunodeppressive known pathological conditions was excluded, as well as any patient with a pathological report describing a normal appendix.
* Patients were divided into four groups according to the interval of time calculated from the onset of symptoms to diagnostic: Group I from 0 to 24 h, Group II from 25 to 48 h, Group III from 49 to 72 h and Group IV more than 73 h.
* At admission demographic, clinical data, and the interval of time from the onset of symptoms to diagnostic was recorded, together with the White Blood Cell (WBC) count, C-reactive protein (CRP) values, and SIRS score.
* The primary outcome measure was to determine the expected systemic inflammatory response to acute appendicitis according to established groups of time intervals from the onset of symptoms to diagnostic using the SIRS for that purpose.
* The secondary outcome measure was the analysis of the CRP to measure the systemic inflammatory response, as another parameter which is habitually included within the diagnostic study of patients with suspected appendicitis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with appendicitis

Exclusion Criteria:

* Any patient with immunosuppressive or immunodeppressive known pathological conditions
* Any patient with a pathological report describing a normal appendix

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with appendicitis operated on and confirmed with biopsy
Sampling Method: Non-Probability Sample
Enrollment: 183 (Actual)
Dates: Start 2011-01; Primary Completion 2012-01 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
THE EXPECTED SYSTEMIC INFLAMMATORY RESPONSE TO APPENDICITIS | 0 to more than 72 hours
  Four groups of time intervals divided as follows:
  Group I: 0 - 24 hours Group II: 25 - 48 hours Group III: 49 - 72 hours Group IV: More than 73 hours

SECONDARY OUTCOMES:
THE ANALYSIS OF C REACTIVE PROTEIN TO MEASURE THE SYSTEMIC INFLAMMATORY RESPONSE TO APPENDICITIS | from 0 to more than 72 hours
  Measurements of C-reactive protein levels

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo A Beltran, M.D., Principal Investigator — La Serena Hospital
Locations (1):
- Hospital de La Serena (La Serena Hospital), La Serena, Coquimbo Region, Chile